CLINICAL TRIAL: NCT01499290
Title: A Phase III, Randomized, Multicenter, Double Blind, Double-Dummy, Parallel-Group, Comparative Study to Determine the Efficacy, Safety, and Tolerability of Ceftazidime Avibactam Plus Metronidazole Versus Meropenem in the Treatment of Complicated Intra-Abdominal Infections In Hospitalized Adults
Brief Title: Compare Ceftazidime-Avibactam + Metronidazole Versus Meropenem for Hospitalized Adults With Complicated Intra-Abdominal Infections
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D4280C00001; 2011-003893-97; NCT01500239 (obsolete NCT alias)
Record Dates: First submitted 2011-12-19; First posted 2011-12-26 (Estimated); Results first posted 2016-03-01 (Estimated); Last update posted 2017-09-06 (Actual); Status verified 2017-08

CONDITIONS: Complicated Intra-Abdominal Infection
Keywords: Ceftazidime; Meropenem; Metronidazole; Anti-Bacterial Agents; Anti-Infective Agents; Antiprotozoal Agents; Antiparasitic Agents; cIAI, Complicated Intra-Abdominal Infection
MeSH Terms: interventions — Metronidazole; Meropenem

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- CAZ-AVI + Metronidazole (Experimental): IV treatment
  Interventions: Drug: CAZ-AVI; Drug: Metronidazole
- Meropenem (Active Comparator): IV treatment
  Interventions: Drug: Meropenem

INTERVENTIONS:
Drug: CAZ-AVI — Ceftazidime 2000 mg and 500 mg of avibactam
  Arms: CAZ-AVI + Metronidazole
Drug: Metronidazole — 500 mg of Metronidazole
  Arms: CAZ-AVI + Metronidazole
Drug: Meropenem — 1 gram of Meropenem
  Arms: Meropenem

SUMMARY:
The purpose of this study is to evaluate the effects of Ceftazidime Avibactam plus Metronidazole compared to Meropenem for treating hospitalized patients with complicated intra-abdominal infections.

DETAILED DESCRIPTION:
A Phase III, Randomized, Multicenter, Double Blind, Double-Dummy, Parallel-Group, Comparative Study to Determine the Efficacy, Safety, and Tolerability of Ceftazidime Avibactam Plus Metronidazole Versus Meropenem in the Treatment of Complicated Intra-Abdominal Infections In Hospitalized Adults

ELIGIBILITY:
Inclusion Criteria:

* 18 to 90 years of age inclusive
* Female patient is authorized to participate if at least one of the following criteria are met:

  1. Surgical sterilization
  2. Age ≥50 years and postmenopausal as defined by amenorrhea for 12 months or more following cessation of all exogenous hormonal treatments
  3. Age <50 years and postmenopausal as defined by documented LH and FSH levels in the postmenopausal range PLUS amenorrhea for 12 months or more following cessation of all exogenous hormonal treatments
  4. Patient has a negative serum pregnancy test (serum ß-human chorionic gonadotropin [ß-hCG]) within 1 day prior to study entry, and agrees to use highly effective contraception methods during treatment and for at least 7 days after last dose of IV study therapy
* Intraoperative/postoperative enrollment with confirmation (presence of pus within the abdominal cavity) of an intra-abdominal infection associated with peritonitis
* Confirmation of infection by surgical intervention within 24 hours of entry: evidence of systemic inflammatory response; physical findings consistent with intra-abdominal infection; supportive radiologic imaging findings of intra-abdominal infections

Exclusion Criteria:

* Patient is diagnosed with traumatic bowel perforation undergoing surgery within 12 hours; perforation of gastroduodenal ulcers undergoing surgery within 24 hours. Other intra-abdominal processes in which primary etiology is not likely to be infectious
* Patient has abdominal wall abscess or bowel obstruction without perforation or ischemic bowel without perforation
* Patient has suspected intra-abdominal infections due to fungus, parasites, virus or tuberculosis
* Patient is considered unlikely to survive the 6 to 8 week study period or has a rapidly progressive or terminal illness, including septic shock that is associated with a high risk of mortality

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 493 (Actual)
Dates: Start 2012-03; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Newell, MBBS, MRCP, Study Director — AstraZeneca
Locations (56):
- United States (4):
  - Research Site, Chula Vista, California
  - Research Site, San Diego, California
  - Research Site, St Louis, Missouri
  - Research Site, Somers Point, New Jersey
- Argentina (2):
  - Research Site, Córdoba
  - Research Site, Rosario
- Bulgaria (2):
  - Research Site, Rousse
  - Research Site, Varna
- Research Site, Zagreb, Croatia
- Czechia (6):
  - Research Site, Děčín
  - Research Site, Hradec Králové
  - Research Site, Jihlava
  - Research Site, Olomouc
  - Research Site, Prague
  - Research Site, Teplice
- Hungary (2):
  - Research Site, Budapest
  - Research Site, Székesfehérvár
- India (4):
  - Research Site, Bangalore
  - Research Site, Pune
  - Research Site, Trivandrum
  - Research Site, Vadodara
- Israel (2):
  - Research Site, Hadera
  - Research Site, Haifa
- Research Site, Riga, Latvia
- Research Site, Alor Star, Malaysia
- Mexico (3):
  - Research Site, Durango
  - Research Site, Guadalajara, Jalisco
  - Research Site, Mexico City
- Netherlands (2):
  - Research Site, 's-Hertogenbosch
  - Research Site, Enschede
- Peru (4):
  - Research Site, Arequipa
  - Research Site, Cercardo de Lima
  - Research Site, Lima
  - Research Site, Trujillo
- Romania (2):
  - Research Site, Cluj-Napoca
  - Research Site, Iași
- Russia (4):
  - Research Site, Kemerovo
  - Research Site, Moscow
  - Research Site, Saratov
  - Research Site, Vsevolozhsk
- Research Site, Pretoria, South Africa
- Spain (3):
  - Research Site, Alcorcón
  - Research Site, Elche
  - Research Site, Sabadell(Barcelona)
- Taiwan (4):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
- Thailand (3):
  - Research Site, Bangkok
  - Research Site, Khon Kaen
  - Research Site, Phisanulok
- Ukraine (5):
  - Research Site, Dnipropetrovsk
  - Research Site, Ivano-Frankivsk
  - Research Site, Kharkiv
  - Research Site, Kyiv
  - Research Site, Zaporizhzhya

REFERENCES:
- [Background] Mazuski JE, Gasink LB, Armstrong J, Broadhurst H, Stone GG, Rank D, Llorens L, Newell P, Pachl J. Efficacy and Safety of Ceftazidime-Avibactam Plus Metronidazole Versus Meropenem in the Treatment of Complicated Intra-abdominal Infection: Results From a Randomized, Controlled, Double-Blind, Phase 3 Program. Clin Infect Dis. 2016 Jun 1;62(11):1380-1389. doi: 10.1093/cid/ciw133. Epub 2016 Mar 8. PMID 26962078
- [Derived] Torres A, Wible M, Tawadrous M, Irani P, Stone GG, Quintana A, Debabov D, Burroughs M, Bradford PA, Kollef M. Efficacy and safety of ceftazidime/avibactam in patients with infections caused by beta-lactamase-producing Gram-negative pathogens: a pooled analysis from the Phase 3 clinical trial programme. J Antimicrob Chemother. 2023 Nov 6;78(11):2672-2682. doi: 10.1093/jac/dkad280. PMID 37700689
- [Derived] Cheng K, Newell P, Chow JW, Broadhurst H, Wilson D, Yates K, Wardman A. Safety Profile of Ceftazidime-Avibactam: Pooled Data from the Adult Phase II and Phase III Clinical Trial Programme. Drug Saf. 2020 Aug;43(8):751-766. doi: 10.1007/s40264-020-00934-3. PMID 32602065
- [Derived] Kongnakorn T, Eckmann C, Bassetti M, Tichy E, Di Virgilio R, Baillon-Plot N, Charbonneau C. Cost-effectiveness analysis comparing ceftazidime/avibactam (CAZ-AVI) as empirical treatment comparing to ceftolozane/tazobactam and to meropenem for complicated intra-abdominal infection (cIAI). Antimicrob Resist Infect Control. 2019 Dec 21;8:204. doi: 10.1186/s13756-019-0652-x. eCollection 2019. PMID 31890160
- [Derived] Li J, Lovern M, Green ML, Chiu J, Zhou D, Comisar C, Xiong Y, Hing J, MacPherson M, Wright JG, Riccobene T, Carrothers TJ, Das S. Ceftazidime-Avibactam Population Pharmacokinetic Modeling and Pharmacodynamic Target Attainment Across Adult Indications and Patient Subgroups. Clin Transl Sci. 2019 Mar;12(2):151-163. doi: 10.1111/cts.12585. Epub 2018 Sep 28. PMID 30221827
- [Derived] Nichols WW, Stone GG, Newell P, Broadhurst H, Wardman A, MacPherson M, Yates K, Riccobene T, Critchley IA, Das S. Ceftazidime-Avibactam Susceptibility Breakpoints against Enterobacteriaceae and Pseudomonas aeruginosa. Antimicrob Agents Chemother. 2018 Oct 24;62(11):e02590-17. doi: 10.1128/AAC.02590-17. Print 2018 Nov. PMID 30061279
- [Derived] Stone GG, Newell P, Gasink LB, Broadhurst H, Wardman A, Yates K, Chen Z, Song J, Chow JW. Clinical activity of ceftazidime/avibactam against MDR Enterobacteriaceae and Pseudomonas aeruginosa: pooled data from the ceftazidime/avibactam Phase III clinical trial programme. J Antimicrob Chemother. 2018 Sep 1;73(9):2519-2523. doi: 10.1093/jac/dky204. PMID 29912399
- [Derived] Stone GG, Newell P, Bradford PA. In Vitro Activity of Ceftazidime-Avibactam against Isolates from Patients in a Phase 3 Clinical Trial for Treatment of Complicated Intra-abdominal Infections. Antimicrob Agents Chemother. 2018 Jun 26;62(7):e02584-17. doi: 10.1128/AAC.02584-17. Print 2018 Jul. PMID 29686147
- [Derived] Mendes RE, Castanheira M, Woosley LN, Stone GG, Bradford PA, Flamm RK. Molecular beta-Lactamase Characterization of Aerobic Gram-Negative Pathogens Recovered from Patients Enrolled in the Ceftazidime-Avibactam Phase 3 Trials for Complicated Intra-abdominal Infections, with Efficacies Analyzed against Susceptible and Resistant Subsets. Antimicrob Agents Chemother. 2017 May 24;61(6):e02447-16. doi: 10.1128/AAC.02447-16. Print 2017 Jun. PMID 28348155
- Available data/document: Study Protocol: D4280C00001 Revised CSP — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1448&filename=RECLAIM%201%20(D4280C00001)%20Protocol.pdf — RECLAIM 1 (D4280C00001) Revised Clinical Study Protocol

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Results from two identical protocols D4280C00001 and D4280C00005 combined into a single database with agreement from FDA and EMA. First patient enrolled 22 March 2012 and last patient's last visit was 07 April 2014. Patients were adults hospitalised with complicated intra-abdominal infection (cIAI) that required surgery and IV antibiotics.
Pre-assignment Details: After obtaining written informed consent patients underwent a preliminary evaluation for eligibility within the 24-hour period prior to initiation of IV study therapy. eligible patients were randomized to 1 of 2 treatment groups in a 1:1 ratio according to the central randomization schedule.
Groups:
- CAZ-AVI + Metronidazole: CAZ (2000mg)/AVI (500mg): IV treatment
- Meropenem: 1000 mg: IV treatment
Period: Overall Study
Arm/Group | CAZ-AVI + Metronidazole | Meropenem
Started | 529 (Patients dosed in pooled protocols D4280C00001/D4280C00005 (NCT01499290/NCT01500239) agreed with FDA) | 529 (Patients dosed in pooled protocols D4280C00001/D4280C00005 (NCT01499290/NCT01500239) agreed with FDA)
Completed | 474 ((Numbers indicate patients who completed treatment)) | 494 ((Numbers indicate patients who completed treatment))
Not Completed | 55 | 35
Not completed — Withdrawal by Subject | 22 | 15
Not completed — Not specified in study report | 11 | 5
Not completed — Condition improved/subject recovered | 1 | 0
Not completed — Lack of Efficacy | 7 | 8
Not completed — Adverse Event | 14 | 7

BASELINE CHARACTERISTICS:
Population: The MITT analysis set includes all patients who met the disease definition for cIAI and received at least 1 dose of study drug. 15 patients excluded received at least one dose of study drug but failed the minimum disease criteria.
Groups:
- Total: Total of all reporting groups
Arm/Group | CAZ-AVI + Metronidazole | Meropenem | Total
Number analyzed (Participants) | 520 | 523 | 1043
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.8 (17.48) | 50.3 (18.29) | 50.0 (17.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 194 | 191 | 385
  Male | 326 | 332 | 658

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response at the Test of Cure (TOC) Visit in the Microbiologically Modified Intent-To-Treat (mMITT) Analysis Set (Primary Outcome for FDA).
Description: The number of patients meeting the cure criteria: complete resolution or significant improvement of signs and symptoms of the index infection such that no further antibacterial therapy, drainage, or surgical intervention is necessary. Indeterminate response are where study data were not available for evaluation of efficacy for any reason, including patient lost to follow-up or assessment not undertaken such that a determination of clinical response could not be made, death where cIAI was clearly noncontributory or circumstances that precluded classification as a cure or failure. Results from two identical protocols D4280C00001 and D4280C00005 combined into a single database with agreement from FDA and EMA.
Time Frame: TOC: 28 to 35 days after start of study drug
Population: The mMITT analysis set included all randomized patients who met the disease definition of cIAI and had at least 1 etiologic pathogen identified at study entry (regardless of isolate susceptibilities). Patients with a bacterial species typically not expected to respond to both study drugs were excluded.
Measure: Number; unit: Participants
Arm/Group | CAZ-AVI + Metronidazole | Meropenem
Number analyzed (Participants) | 413 | 410
Participants
  Clinical cure | 337 | 349
  Clinical failure | 37 | 30
  Indeterminate | 39 | 31
Statistical Analysis 1: Comparison: CAZ-AVI + Metronidazole vs Meropenem; The primary objective of this study (FDA agreed) was to determine the noninferiority in the clinical cure rate for CAZ-AVI compared to that for Meropenem at TOC in the mMITT in adult subjects with cIAI; Test type: Non-Inferiority or Equivalence — Non-inferiority was determined by comparing the lower limit of the 95% confidence interval for risk difference (corresponding to a 97.5% 1-sided lower bound) to the non-inferiority marging of -12.5%; Risk Difference (RD) = -3.5, 95% CI 2-sided [-8.64 to 1.58]

2. Primary Outcome: Clinical Response at the TOC Visit in the Modified Intent-To-Treat Analysis Set (Co-primary Outcome for Rest of World [ROW]).
Description: The number of patients meeting the cure criteria: complete resolution or significant improvement of signs and symptoms of the index infection such that no further antibacterial therapy, drainage, or surgical intervention was necessary. Indeterminate response are where study data were not available for evaluation of efficacy for any reason, including patient lost to follow-up or assessment not undertaken such that a determination of clinical response could not be made, dDeath where cIAI was clearly noncontributory or circumstances that precluded classification as a cure or failure.
Time Frame: TOC: 28 to 35 days after start of study drug
Population: The MITT analysis set included all randomized patients who met the disease definition of cIAI and who received any amount of study drug.
Measure: Number; unit: Participants
Arm/Group | CAZ-AVI + Metronidazole | Meropenem
Number analyzed (Participants) | 520 | 523
Participants
  Clinical cure | 429 | 444
  Clinical failure | 47 | 39
  Indeterminate | 44 | 40
Statistical Analysis 1: Comparison: CAZ-AVI + Metronidazole vs Meropenem; The co-primary objective of this study (ROW agreed) was to determine the noninferiority in the clinical cure rate for CAZ-AVI compared to that for Meropenem at TOC in the MITT in adult subjects with cIAI; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Risk Difference (RD) = -2.4, 95% CI 2-sided [-6.90 to 2.10]

3. Primary Outcome: Clinical Response at the TOC Visit in the Clinically Evaulable (CE) Analysis Set (Co-primary Outcome for Rest of World [ROW]).
Description: The number of patients meeting the cure criteria: complete resolution or significant improvement of signs and symptoms of the index infection such that no further antibacterial therapy, drainage, or surgical intervention was necessary.
Time Frame: TOC: 28 to 35 days after start of study drug
Population: The CE analysis set included all patients who met the disease definition of cIAI and met the stringent criteria for clinical evaluation described in the protocol regarding dosing, concomitant medication, evaluation, etc.
Measure: Number; unit: Participants
Arm/Group | CAZ-AVI + Metronidazole | Meropenem
Number analyzed (Participants) | 410 | 416
Participants
  Clinical cure | 376 | 385
  Clinical failure | 34 | 31
Statistical Analysis 1: Comparison: CAZ-AVI + Metronidazole vs Meropenem; The co-primary objective of this study (ROW agreed) was to determine the noninferiority in the clinical cure rate for CAZ-AVI compared to that for Meropenem at TOC in the CE in adult subjects with cIAI; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Risk Difference (RD) = -0.8, 95% CI 2-sided [-4.61 to 2.89]

4. Secondary Outcome: Clinical Cure at TOC in the Microbiologically Evaluable Analysis Set
Description: as for outcome 3
Time Frame: TOC: 28 to 35 days after start of study drug
Population: ME analysis set defined as all patients included in the CE set with at least 1 Gram negative, aerobic, susceptible pathogen in the initial/prestudy culture.
Measure: Number; unit: Participants
Arm/Group | CAZ-AVI + Metronidazole | Meropenem
Number analyzed (Participants) | 265 | 287
Participants
  Clinical cure | 244 | 272
  Clinical failure | 21 | 15

5. Secondary Outcome: Clinical Cure at TOC in the Extended Microbiologically Evaluable Analysis Set
Description: as for outcome 3
Time Frame: TOC: 28 to 35 days after start of study drug
Population: Extended ME analysis set defined as all patients included in the CE set with at least 1 Gram negative, aerobic, pathogen in the initial/prestudy culture, regardless of susceptibility.
Measure: Number; unit: Participants
Arm/Group | CAZ-AVI + Metronidazole | Meropenem
Number analyzed (Participants) | 270 | 294
Participants
  Clinical cure | 248 | 278
  Clinical failure | 22 | 16

6. Secondary Outcome: Clinical Response by Visit in the Primary Population: Microbiologically Modified Intent-to-Treat (mMITT)
Description: Complete resolution or significant improvement of signs and symptoms of the index infection such that no further antibacterial therapy, drainage, or surgical intervention was necessary. Indeterminate response are where study data were not available for evaluation of efficacy for any reason, including patient lost to follow-up or assessment not undertaken such that a determination of clinical response could not be made, dDeath where cIAI was clearly noncontributory or circumstances that precluded classification as a cure or failure.
Time Frame: EOT: within 24 hours after last dose of study drug. TOC: 28 to 35 days after start of study drug. LFU: 42 to 49 days after start of study drug
Population: as for outcome 1
Measure: Number; unit: Participants
Groups:
- CAZ-AVI + Metronidazole (EOT); Meropenem (EOT): EOT - within 24 hours of last dose of study drug
- CAZ-AVI + Metronidazole (TOC); Meropenem (TOC): TOC - 28 to 35 days after start of study drug
- CAZ-AVI + Metronidazole (LFU); Meropenem (LFU): LFU - 42 to 49 days after start of study drug
Arm/Group | CAZ-AVI + Metronidazole (EOT) | Meropenem (EOT) | CAZ-AVI + Metronidazole (TOC) | Meropenem (TOC) | CAZ-AVI + Metronidazole (LFU) | Meropenem (LFU)
Number analyzed (Participants) | 413 | 410 | 413 | 410 | 413 | 410
Participants
  Clinical cure | 361 | 379 | 337 | 349 | 340 | 347
  Clinical failure | 30 | 19 | 37 | 30 | 38 | 31
  Indeterminate | 22 | 12 | 39 | 31 | 35 | 32

7. Secondary Outcome: Per-patient Microbiological Response in the Microbiologically Modified Intent- To-Treat Analysis Set
Description: Microbiological responses as per the protocoled criteria: responses other than "indeterminate" were classified as "favorable" or "unfavorable." Favorable microbiological response assessments included "eradication" and "presumed eradication." Unfavorable microbiological response assessments included "persistence," "persistence with increasing minimum inhibitory concentration (MIC)," and "presumed persistence." Indeterminate microbiologic response assessments included cases where the clinical response was changed to indeterminate due to a surgical review panel (SRP) assessment of inadequate source control (ie, circumstances that preclude classification as eradication, presumed eradication, persistence, persistence with increasing MIC, and presumed persistence).
Time Frame: EOT: within 24 hours after last dose of study drug. TOC: 28 to 35 days after start of study drug. LFU 42 to 49 days after start of study drug
Population: as for outcome 1
Measure: Number; unit: Participants
Groups:
- CAZ-AVI + Metronidazole (EOT); Meropenem (EOT): EOT - within 24 hours after last dose of study drug
Arm/Group | CAZ-AVI + Metronidazole (EOT) | Meropenem (EOT) | CAZ-AVI + Metronidazole (TOC) | Meropenem (TOC) | CAZ-AVI + Metronidazole (LFU) | Meropenem (LFU)
Number analyzed (Participants) | 413 | 410 | 413 | 410 | 413 | 410
Participants
  Favourable response | 362 | 379 | 337 | 349 | 340 | 347
  Unfavourable response | 30 | 19 | 37 | 31 | 38 | 32
  Indeterminate | 21 | 12 | 39 | 30 | 35 | 31

8. Secondary Outcome: Per-pathogen Microbiological Response at TOC in the Microbiologically Modified Intent-To-Treat Analysis Set.
Description: The number of patients with a favorable per-pathogen microbiological response: favourable microbiological response includes: Eradication Absence of causative pathogen from specimens at the site of infection. Presumed eradication where, repeat cultures were not performed/clinically indicated in a patient who had a clinical response of cure.
Time Frame: TOC: 28 to 35 days after start of study drug.
Population: as for outcome 1
Measure: Number; unit: Participants
Groups:
- CAZ-AVI + Metronidazole: CAZ (2000mg)/AVI (500mg): IV treatment Number of favourable responses
- Meropenem: 1000 mg: IV treatment. Number of favourable responses
- CAZ-AVI + Metronidazole (Denominator): Total number of patiets with each pathogen at baseline (summary only shows pathogens where N>/=10)
- Meropenem (Denominator): Number of patients with pathogen at baseline
Arm/Group | CAZ-AVI + Metronidazole | Meropenem | CAZ-AVI + Metronidazole (Denominator) | Meropenem (Denominator)
Number analyzed (Participants) | 413 | 410 | 413 | 410
Participants
  Citrobacter freundii complex | 14 | 9 | 18 | 12
  Enterobacter aerogenes | 4 | 5 | 5 | 5
  Enterobacter cloacae | 11 | 16 | 13 | 19
  Escherichia coli | 218 | 249 | 271 | 285
  Klebsiella oxytoca | 14 | 12 | 18 | 15
  Klebsiella pneumoniae | 40 | 37 | 51 | 49
  Proteus mirabilis | 5 | 7 | 8 | 9
  Pseudomonas aeruginosa | 30 | 34 | 35 | 36
  Enterococcus avium | 8 | 10 | 8 | 15
  Enterococcus faecalis | 22 | 23 | 31 | 28
  Enterococcus faecium | 13 | 18 | 16 | 22
  Staphylococcus aureus | 17 | 14 | 18 | 14
  Streptococcus anginosus group | 59 | 50 | 72 | 61
  Streptococcus bovis group | 2 | 6 | 3 | 7
  Streptococcus mitis group | 10 | 9 | 15 | 11
  Bacteroides fragilis | 45 | 38 | 52 | 47
  Bacteroides ovatus | 17 | 17 | 22 | 20
  Bacteroides stercoris | 9 | 1 | 10 | 1
  Bacteroides thetaiotaomicron | 18 | 21 | 22 | 25
  Bacteroides uniformis | 4 | 6 | 7 | 7
  Bacteroides vulgatus | 6 | 6 | 8 | 9
  Clostridium perfringens | 7 | 4 | 10 | 4
  Eggerthella lenta | 5 | 7 | 5 | 8
  Parabacteroides distasonis | 13 | 12 | 16 | 13
  Parvimonas micra | 7 | 8 | 7 | 10

9. Secondary Outcome: Clinical Response by Pathogen at TOC for Patients Infected With Ceftazidime-resistant Pathogens in Microbiological Modified Intent to Treat Analysis Set
Description: Complete resolution or significant improvement of signs and symptoms of the index infection such that no further antibacterial therapy, drainage, or surgical intervention was necessary.
Time Frame: Test of Cure: 28 to 35 days after start of study drug
Population: as for outcome 1
Measure: Number; unit: Participants
Groups:
- CAZ-AVI + Metronidazole (Denominator); Meropenem (Denominator): Number of patients with pathogen at baseline
Arm/Group | CAZ-AVI + Metronidazole | Meropenem | CAZ-AVI + Metronidazole (Denominator) | Meropenem (Denominator)
Number analyzed (Participants) | 413 | 410 | 413 | 410
Participants
  All | 39 | 55 | 47 | 64
  Citrobacter freundii complex | 1 | 2 | 1 | 2
  Enterobacter aerogenes | 0 | 1 | 0 | 1
  Enterobacter cloacae | 2 | 7 | 3 | 7
  Escherichia coli | 19 | 31 | 24 | 37
  Klebsiella pneumoniae | 10 | 9 | 13 | 13
  Morganella morganii | 1 | 1 | 2 | 1
  Proteus mirabilis | 2 | 3 | 2 | 3
  Serratia marcescens | 1 | 0 | 1 | 0
  Alcaligenes faecalis | 1 | 2 | 1 | 2
  Comamonas testosteroni | 1 | 0 | 1 | 0
  Pseudomonas aeruginosa | 2 | 4 | 2 | 4

10. Secondary Outcome: Favorable Per-pathogen Microbiological Response for Patients Infected With Ceftazidime-resistant Pathogens in mMITT Analysis Set
Description: as for outcome 8
Time Frame: TOC: 28 to 35 days after start of study drug
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | CAZ-AVI + Metronidazole | Meropenem | CAZ-AVI + Metronidazole (Denominator) | Meropenem (Denominator)
Number analyzed (Participants) | 48 | 64 | 48 | 64
Participants
  Citrobacter freundii complex | 1 | 2 | 2 | 2
  Enterobacter aerogenes | 0 | 1 | 0 | 1
  Enterobacter cloacae | 2 | 7 | 3 | 7
  Escherichia coli | 19 | 31 | 24 | 37
  Klebsiella pneumoniae | 10 | 9 | 13 | 13
  Morganella morganii | 1 | 1 | 2 | 1
  Proteus mirabilis | 2 | 3 | 2 | 3
  Serratia marcescens | 1 | 0 | 1 | 0
  Alcaligenes faecalis | 1 | 2 | 1 | 2
  Comamonas testosteroni | 1 | 0 | 1 | 0
  Pseudomonas aeruginosa | 2 | 4 | 2 | 4

11. Secondary Outcome: Per-patient Microbiological Response at TOC for Patients Infected With Ceftazidime-resistant Pathogens in mMITT Analysis Set
Description: Microbiological responses other than "indeterminate" were classified as "favorable" or "unfavorable." Favorable microbiological response assessments included "eradication" and "presumed eradication." Unfavorable microbiological response assessments included "persistence," "persistence with increasing minimum inhibitory concentration (MIC)," and "presumed persistence." Indeterminate microbiologic response assessments included cases where the clinical response was changed to indeterminate due to an SRP assessment of inadequate source control (ie, circumstances that preclude classification as eradication, presumed eradication, persistence, persistence with increasing MIC, and presumed persistence).
Time Frame: Test of Cure: 28 to 35 days after start of study drug
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | CAZ-AVI + Metronidazole | Meropenem
Number analyzed (Participants) | 48 | 64
Participants
  Favourable | 39 | 55
  Unfavourable | 7 | 1
  indeterminate | 2 | 8

12. Secondary Outcome: Number of Patients Afebrile at Last Observation in the Clinically Evaluable Analysis Set for Patients Who Have Fever at Study Entry
Description: Time to first defervescence was calculated for patients with a fever (>38ºC) at baseline. Defervescence (≤37.8ºC) was defined as the absence of fever based on the highest temperature recorded on each study day.
Time Frame: Test of Cure: 1 to 14 days after start of study drug
Population: Clinically evaluable (CE) with fever, defined as >38ºC at study entry.
Measure: Number; unit: Participants
Arm/Group | CAZ-AVI + Metronidazole | Meropenem
Number analyzed (Participants) | 84 | 78
Participants | 84 | 72

13. Secondary Outcome: Plasma Concentrations for Ceftazidime and Avibactam
Description: Blood samples were taken from all patients on Day 3 for the pharmacokinetic evaluation of ceftazidime and avibactam plasma concentrations
Time Frame: Anytime within 15 minutes prior to or after stopping study drug, anytime between 30 and 90 minutes after stopping study drug, anytime between 300 minutes and 360 minutes after stopping study drug
Population: PK analysis set
Measure: Geometric Mean (Full Range); unit: (NG/ML)
Groups:
- CAZ (1): 30 mins before/after dose
- AVI (1): 30 min before/after dose
- CAZ (2); AVI (2): 30-90 mins after dose
- CAZ (3); AVI (3): 300-360 mins after dose
Arm/Group | CAZ (1) | AVI (1) | CAZ (2) | AVI (2) | CAZ (3) | AVI (3)
Number analyzed (Participants) | 486 | 493 | 484 | 489 | 481 | 484
(NG/ML) | 50823.0 [171 to 3110000] | 9229.4 [13 to 693000] | 40053.1 [155 to 235000] | 7163.9 [15 to 46800] | 10967.6 [159 to 151000] | 1690.7 [14 to 30800]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the screening/consent visit until the late follow-up visit (ie Day -1/0 to Day 42).
Description: AEs spontaneously reported by the patient or care provider or reported in response to the open question from the study center personnel, or revealed by observation were to be collected and recorded in the eCRF.
Arm/Group | CAZ-AVI + Metronidazole | Meropenem
Serious Adverse Events (participants affected / at risk) | 17/529 | 15/529
Other Adverse Events (participants affected / at risk) | 184/529 | 152/529
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CAZ-AVI + Metronidazole (N=529) | Meropenem (N=529)
Myocardial infarction (Cardiac disorders) | 1 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Renal failure acute (Renal and urinary disorders) | 5 | 0
Transaminases increased (Investigations) | 0 | 2
Gastrointestinal stoma necrosis (Injury, poisoning and procedural complications) | 2 | 0
Abdominal abscess (Infections and infestations) | 0 | 2
Bronchopneumonia (Infections and infestations) | 2 | 2
Candida sepsis (Infections and infestations) | 2 | 0
Cardiac failure (Cardiac disorders) | 2 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 2
Colonic abscess (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0
Empyema (Infections and infestations) | 1 | 0
Enterococcal bacteraemia (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 0 | 1
Septic enceohalopathy (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 0 | 1
Systematic candida (Infections and infestations) | 0 | 1
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Delirium tremens (Psychiatric disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1
Polyneuropathy (Nervous system disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Left ventricular failure (Cardiac disorders) | 1 | 0
Right ventricular failure (Cardiac disorders) | 1 | 0
Shock (Vascular disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Colonic fistula (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal hypomotility (Gastrointestinal disorders) | 1 | 0
Ileal perforation (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 1 | 0
Localised intraabdominal fluid collection (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Small intestine perforation (Gastrointestinal disorders) | 1 | 0
Subileus (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Volvulus (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Bile duct obstruction (Hepatobiliary disorders) | 1 | 1
Biloma (Hepatobiliary disorders) | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1
Critical illness myopathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Multi-organ failure (General disorders) | 1 | 0
Sudden death (General disorders) | 1 | 1
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 1 | 1
Anastomotic leak (Injury, poisoning and procedural complications) | 1 | 0
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 1 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 1
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 1 | 0
Post procedural bile leak (Injury, poisoning and procedural complications) | 0 | 1
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Suture related complication (Injury, poisoning and procedural complications) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Wound evisceration (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CAZ-AVI + Metronidazole (N=529) | Meropenem (N=529)
Wound infection (Infections and infestations) | 13 | 11
Headache (Nervous system disorders) | 15 | 9
Hypertension (Vascular disorders) | 15 | 24
Hypotension (Vascular disorders) | 12 | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 13
Diarrhoea (Gastrointestinal disorders) | 40 | 17
Nausea (Gastrointestinal disorders) | 36 | 24
Vomiting (Gastrointestinal disorders) | 24 | 10
Constipation (Gastrointestinal disorders) | 8 | 20
Pyrexia (General disorders) | 24 | 24
Asthenia (General disorders) | 10 | 12
Abdominal distension (Gastrointestinal disorders) | 10 | 11
Phlebitis (Vascular disorders) | 10 | 11
Anaemia (Blood and lymphatic system disorders) | 11 | 9

LIMITATIONS AND CAVEATS:
This summary describes data collected from two identical CSPs (D4280C00001 and D4280C00005). With agreement from the EMA and the FDA the data have been combined into a single study database.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI shall not publish results until the earliest of (i) date of the 1st study publication (joint between PI, sponsor and study sites) (ii) 18 months after study completion, or (iii) sponsor notification that no multi-center publication is to be made. The PI submits the publication for review 60 days before submission. Sponsor may embargo for a further 90 days to protect IP rights. Sponsor may request removal of confidential and/or proprietry information.